CLINICAL TRIAL: NCT07382882
Title: Wpływ Podawanego Doustnie Ekstraktu z Aronii, Jagody Kamczackiej Oraz Czarnej Jagody na Stan narządu Wzroku.
Brief Title: The Effect of Orally Administered Extracts of Chokeberry, Kamchatka Berry and Blueberry on the Condition of the Eye.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Dorota Szumny, Principal Investigator, Wroclaw Medical University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: KB 672/2022, KB 258/2025; SUBZ.A080.22.076 and Subz.A080 (Other Grant/Funding Number: Wroclaw Medical University)
Record Dates: First submitted 2026-01-14; First posted 2026-02-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Presbyopia
Keywords: Presbyopia; iridoids; anthocyanins; chokeberry; blueberry; honeysuckle berry
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Intervention Model Description: randomised, double-blind, placebo-controlled, two-period crossover trial
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention 1: Dietary Supplement: AKB (Experimental): dose: 400 mg capsule, 1 capsule BID (2×/d) throug 6 weeks
  Interventions: Dietary Supplement: AKB
- Intervention 2: Placebo (Placebo Comparator): maltodextrin + natural caramel colouring, BID, 6 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: AKB — Standardized berry extract (Aronia melanocarpa, Lonicera caerulea, Vaccinium myrtillus), 400 mg capsule, BID, 6 weeks
  Arms: Intervention 1: Dietary Supplement: AKB
Other: Placebo — Matching placebo capsules (maltodextrin + colouring), BID, 6 weeks
  Arms: Intervention 2: Placebo

SUMMARY:
This study evaluated whether a standardized berry-extract dietary supplement (AKB; Aronia melanocarpa, Lonicera caerulea, Vaccinium myrtillus) improves visual function in adults with presbyopia. In a randomized, double-blind, placebo-controlled two-period crossover design, participants received AKB 400 mg twice daily and placebo for 6 weeks each, separated by a 5-week washout. Visual function and retinal/neuronal measures were assessed with contrast sensitivity testing, visual fields, VEP, and OCT/AngioOCT. Serum biomarkers related to lens and retinal physiology were also measured.

DETAILED DESCRIPTION:
Participants were randomized to one of two sequences (AKB→placebo or placebo→AKB). Each treatment period lasted 6 weeks, separated by a 5-week washout. Ophthalmological assessments were performed at baseline and during the final week of each treatment period. The primary analysis compared within-participant changes after AKB versus placebo.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 50 years.

Clinical diagnosis of presbyopia.

Best-corrected visual acuity (BCVA) ≥ 20/40.

Spherical refraction between -3.0 and +3.0 diopters (D).

Cylinder correction ≤ ±3.0 D.

Exclusion Criteria:

Age < 50 years.

History of ocular surgery within 12 months prior to enrollment.

Presence of ocular diseases/conditions that may affect outcomes, including:

Macular degeneration

Diabetic retinopathy

Retinal vein occlusion

Glaucoma

Other significant acquired or hereditary eye conditions

Neurological disorders affecting visual fields.

Refractive error outside eligibility limits:

Spherical refraction < -3.0 D or > +3.0 D

Cylinder correction > ±3.0 D

Systemic conditions that may influence optic nerve head perfusion, including:

Hypotension

Severe circulatory failure

Vascular endothelial disorders

Gastrointestinal conditions, including:

Hyperacidity

Peptic ulcer disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Change in visual field (automated perimetry) | Baseline and Week 6.
  Change from baseline in visual field mean deviation (MD, dB) measured by standard automated perimetry measured by Humphrey Field Analyzer.
Change in PVEP P100 latency (pattern size 1.0) | Baseline and Week 6.
  Change from baseline to Week 6 in PVEP P100 latency (ms) measured by pattern-reversal VEP (pattern size 1.0).
Change in PVEP P100 amplitude (pattern size 1.0) | Baseline and Week 6.
  Change from baseline to Week 6 in PVEP P100 amplitude (µV) measured by pattern-reversal VEP (pattern size 1.0).
Change in PVEP P100 latency (pattern size 0.3) | Baseline and Week 6.
  Change from baseline to Week 6 in PVEP P100 latency (ms) measured by pattern-reversal VEP (pattern size 0.3).
Change in PVEP P100 amplitude (pattern size 0.3) | Baseline and Week 6.
  Change from baseline to Week 6 in PVEP P100 amplitude (µV) measured by pattern-reversal VEP (pattern size 0.3).
Change in OCT / OCT-angiography parameters | Baseline and Week 6.
  Change from baseline in RNFL thickness (µm) measured by spectral-domain OCT.
Change in OCT / OCT-angiography parameters | Baseline and Week 6.
  Change from baseline in central macular thickness (µm) measured by spectral-domain OCT.
Change in OCT / OCT-angiography parameters | Baseline and Week 6.
  Change from baseline in GCC thickness (µm) measured by spectral-domain OCT.
Change in OCT / OCT-angiography parameters | Baseline and Week 6.
  Change from baseline in retinal vessel density (%) measured by OCT-angiography.

SECONDARY OUTCOMES:
Change in serum CRYAA concentration | One month.
  Change from baseline in serum CRYAA concentration measured by ELISA (ng/mL).
Change in serum CRYAB concentration | one month
  Change from baseline in serum CRYAB concentration measured by ELISA (ng/mL).
Change in serum TRPV4 level | one month
  Change from baseline in serum TRPV4 level measured by ELISA (ng/mL).

CONTACTS AND LOCATIONS:
Locations (1):
- Wroclaw Medical University, Wroclaw, Poland